CLINICAL TRIAL: NCT01363297
Title: An Open-label, Phase 1/2 Study Of Inotuzumab Ozogamicin In Subjects With Relapsed Or Refractory Cd22-positive Acute Lymphocytic Leukemia
Brief Title: Study Evaluating Inotuzumab Ozogamicin In Acute Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: UCB Pharma (Industry)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: B1931010; 3129K6-1106 (Other: Alias Study Number)
Record Dates: First submitted 2011-05-11; First posted 2011-06-01 (Estimated); Results first posted 2017-04-13 (Actual); Last update posted 2017-04-13 (Actual); Status verified 2017-03

CONDITIONS: Acute Lymphocytic Leukemia
Keywords: Relapsed/Refractory Acute Lymphocytic Leukemia (ALL)
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Inotuzumab Ozogamicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Inotuzumab Ozogamicin (Experimental)
  Interventions: Drug: Inotuzumab Ozogamicin

INTERVENTIONS:
Drug: Inotuzumab Ozogamicin — Part 1: Administered intravenously as 2 - 3 weekly doses over a 28-day cycle for a maximum of 6 cycles. Total dose per cycle 0.8 mg/m^2 to 2.0 mg/m^2.
  Part 2 Expansion and Part 3 Phase 2: Administered intravenously as 3 weekly doses over a 28-day cycle for a maximum of 6 cycles. Total initial dose per cycle 1.8 mg/m^2.
  Other Names: CMC-544

SUMMARY:
The Phase 1 portion of this study will assess the safety, tolerability and efficacy at increasing dose levels of inotuzumab ozogamicin in subjects with CD22-positive relapsed or refractory adult acute lymphocytic leukemia (ALL) in order to select the recommended phase 2 dose (RP2D) and schedule. The Phase 2 portion of the study will evaluate the efficacy of inotuzumab ozogamicin as measured by hematologic remission rate (CR + CRi) in patients in second or later salvage status.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with CD22-positive ALL with either refractory disease (i.e. disease progression or no response while receiving their most recent prior anti-cancer therapy), or relapsed disease (i.e. response to their most recent prior anti-cancer therapy with subsequent relapse). Subjects enrolled in the Phase 2 portion of the study must be due to receive salvage 2 or later therapy.
* Subjects with Philadelphia chromosome-positive (Ph+) ALL must have failed standard treatment with at least one tyrosine kinase inhibitor.
* Adequate renal and hepatic function, and negative pregnancy test for women of childbearing potential.

Exclusion Criteria:

* Subjects with isolated extramedullary relapse or active central nervous system (CNS) leukemia.
* Prior allogeneic hematopoietic stem cell transplant (HSCT) or other anti-CD22 immunotherapy within 4 months, or active graft versus host disease (GvHD) at study entry.
* Evidence or history of veno-occlusive disease (VOD) or sinusoidal obstruction syndrome (SOS).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2011-08; Primary Completion 2014-08 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (15):
- United States (15):
  - City of Hope National Medical Center, Duarte, California
  - Stanford Unversity Cancer Clinical Trials Office, Palo Alto, California
  - Stanford Unversity Hospital and Clinics, CTRU, Palo Alto, California
  - Stanford Cancer Institute, Stanford, California
  - Stanford University Hospital and Clinics, Stanford, California
  - The University of Chicago Medical Center, Chicago, Illinois
  - Massachusetts General Hospital (MGH), Boston, Massachusetts
  - Brigham and Women's Hospital (BWH), Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Karmanos Cancer Institute at Farmington Hills, Farmington Hills, Michigan
  - Cleveland Clinic, Cleveland, Ohio
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Seattle Cancer Care Alliance, Seattle, Washington

REFERENCES:
- [Derived] Shi Z, Zhu Y, Zhang J, Chen B. Monoclonal antibodies: new chance in the management of B-cell acute lymphoblastic leukemia. Hematology. 2022 Dec;27(1):642-652. doi: 10.1080/16078454.2022.2074704. PMID 35622074
- [Derived] Stock W, Martinelli G, Stelljes M, DeAngelo DJ, Gokbuget N, Advani AS, O'Brien S, Liedtke M, Merchant AA, Cassaday RD, Wang T, Zhang H, Vandendries E, Jabbour E, Marks DI, Kantarjian HM. Efficacy of inotuzumab ozogamicin in patients with Philadelphia chromosome-positive relapsed/refractory acute lymphoblastic leukemia. Cancer. 2021 Mar 15;127(6):905-913. doi: 10.1002/cncr.33321. Epub 2020 Nov 24. PMID 33231879
- [Derived] DeAngelo DJ, Stock W, Stein AS, Shustov A, Liedtke M, Schiffer CA, Vandendries E, Liau K, Ananthakrishnan R, Boni J, Laird AD, Fostvedt L, Kantarjian HM, Advani AS. Inotuzumab ozogamicin in adults with relapsed or refractory CD22-positive acute lymphoblastic leukemia: a phase 1/2 study. Blood Adv. 2017 Jun 27;1(15):1167-1180. doi: 10.1182/bloodadvances.2016001925. eCollection 2017 Jun 27. PMID 29296758
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1931010&StudyName=Study%20Evaluating%20Inotuzumab%20Ozogamicin%20In%20Acute%20Lymphocytic%20Leukemia

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1 - Dose-Finding: IV Inotuzumab Ozogamicin 1.2 mg/m^2: IV inotuzumab ozogamicin 1.2 mg/m^2 given in 2 doses over a 28-day cycle (0.8 mg/m^2 on Day 1 and 0.4 mg/m^2 on Day 15) for a maximum of 6 cycles
- Phase 1 - Dose-Finding: IV Inotuzumab Ozogamicin 1.6 mg/m^2: IV inotuzumab ozogamicin 1.6 mg/m^2 given in 3 doses over a 28-day cycle (0.8 mg/m^2 on Day 1 and 0.4 mg/m^2 on Days 8 and 15) for a maximum of 6 cycles
- Phase 1 - Dose-Finding: IV Inotuzumab Ozogamicin 1.8 mg/m^2; Phase 1 - Expansion Phase: IV Inotuzumab Ozogamicin 1.8 mg/m^2; Phase 2: IV Inotuzumab Ozogamicin 1.8mg/m^2: IV inotuzumab ozogamicin 1.8 mg/m^2 given in 3 doses over a 28-day cycle (0.8 mg/m^2 on Day 1 and 0.5 mg/m^2 on Days 8 and 15) for a maximum of 6 cycles
Period: Overall Study
Arm/Group | Phase 1 - Dose-Finding: IV Inotuzumab Ozogamicin 1.2 mg/m^2 | Phase 1 - Dose-Finding: IV Inotuzumab Ozogamicin 1.6 mg/m^2 | Phase 1 - Dose-Finding: IV Inotuzumab Ozogamicin 1.8 mg/m^2 | Phase 1 - Expansion Phase: IV Inotuzumab Ozogamicin 1.8 mg/m^2 | Phase 2: IV Inotuzumab Ozogamicin 1.8mg/m^2
Started | 3 | 12 | 9 | 13 | 35
Completed | 0 | 6 | 3 | 3 | 4
Not Completed | 3 | 6 | 6 | 10 | 31
Not completed — Other | 0 | 0 | 0 | 0 | 1
Not completed — Death | 3 | 6 | 6 | 10 | 30

BASELINE CHARACTERISTICS:
Population: Safety analysis set - included all enrolled participants who received at least 1 dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1 - Dose-Finding: IV Inotuzumab Ozogamicin 1.2 mg/m^2 | Phase 1 - Dose-Finding: IV Inotuzumab Ozogamicin 1.6 mg/m^2 | Phase 1 - Dose-Finding: IV Inotuzumab Ozogamicin 1.8 mg/m^2 | Phase 1 - Expansion Phase: IV Inotuzumab Ozogamicin 1.8 mg/m^2 | Phase 2: IV Inotuzumab Ozogamicin 1.8mg/m^2 | Total
Number analyzed (Participants) | 3 | 12 | 9 | 13 | 35 | 72
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.7 (1.53) | 44.9 (18.06) | 43.1 (18.37) | 53.4 (13.82) | 40.7 (17.08) | 44.9 (17.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 6 | 6 | 8 | 21
  Male | 3 | 11 | 3 | 7 | 27 | 51

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Reporting Dose Limiting Toxicities (DLTs) During the Phase 1 Dose-Finding Phase
Description: DLT was any of the following in the first cycle & attributable to inotuzumab ozogamicin: any greater than or equal to (≥) Grade 4 non-hematologic toxicity except nausea/vomiting (if manageable with supportive care), alopecia, & toxicities secondary to neutropenia & sepsis; prolonged myelosuppression (absolute neutrophil count [ANC] less than [<] 500 per microliter [/µL] or platelet count <25,000/µL in bone marrow with <5 percent (%) blasts & no evidence of leukemia more than 45 days beyond the most recent dose of test article); any Grade 3 non-hematologic toxicity (excluding toxicities such as alopecia or those secondary to neutropenia & sepsis) not resolving to ≥ Grade 2 within 7 days of the most recent dose of test article or was clinically significant irrespective of duration; any ≥ Grade 3 elevation of alanine aminotransferase, aspartate aminotransferase or bilirubin lasting ≥7 days; any test article related toxicity resulting in permanent discontinuation of test article.
Time Frame: Cycle 1
Population: Safety analysis set
Measure: Number; unit: Percentage of Participants
Groups:
- Phase 1 - Dose Finding: IV Inotuzumab Ozogamicin 1.6 mg/m^2: IV inotuzumab ozogamicin 1.6 mg/m^2 given in 3 doses over a 28-day cycle (0.8 mg/m^2 on Day 1 and 0.4 mg/m^2 on Days 8 and 15) for a maximum of 6 cycles
Arm/Group | Phase 1 - Dose-Finding: IV Inotuzumab Ozogamicin 1.2 mg/m^2 | Phase 1 - Dose Finding: IV Inotuzumab Ozogamicin 1.6 mg/m^2 | Phase 1 - Dose-Finding: IV Inotuzumab Ozogamicin 1.8 mg/m^2
Number analyzed (Participants) | 3 | 12 | 9
Percentage of Participants | 0 | 0 | 11.1

2. Primary Outcome: Percentage of Participants With Preliminary Satisfactory Response (Complete Response [CR], CR With Incomplete Count Recovery [CRi], Partial Response [PR], or Resistant Disease [RD]) Indicating Disease Stability After First Dose During Phase 1 Dose-Finding
Description: CR was the disappearance of leukemia indicated by <5% marrow blasts and absence of peripheral blood leukemic blasts, with recovery of hematopoiesis defined by ANC ≥1000/µL and platelets ≥100,000/µL. C1 extramedullary disease status was required. CRi was as for CR except with ANC <1000/µL and/or platelets <100,000/µL. PR was an improved or no worsening of acute lymphocytic leukemia indicated by no peripheral blood blasts, and/or at least a 50% decrease in the marrow blast percentage, compared to pre-treatment value, and marrow blast percentage ≥5% and less than or equal to (≤)25% and/or C2 extramedullary disease status. RD occurred if a participant survived ≥7 days following completion of initial treatment course and had persistent leukemia in the most recent peripheral blood smear or bone marrow and/or persistent disease involvement at any extramedullary site after completion of therapy.
Time Frame: From screening to progressive disease or another induction therapy started, up to approximately 2 years
Population: Safety analysis set
Measure: Number; unit: Percentage of Participants
Arm/Group | Phase 1 - Dose-Finding: IV Inotuzumab Ozogamicin 1.2 mg/m^2 | Phase 1 - Dose Finding: IV Inotuzumab Ozogamicin 1.6 mg/m^2 | Phase 1 - Dose-Finding: IV Inotuzumab Ozogamicin 1.8 mg/m^2
Number analyzed (Participants) | 3 | 12 | 9
Percentage of Participants | 100 | 91.7 | 88.9

3. Primary Outcome: Percentage of Participants With CR or CRi During Phase 2
Description: CR was defined as a disappearance of leukemia as indicated by <5% marrow blasts and the absence of peripheral blood leukemic blasts, with recovery of hematopoiesis defined by ANC ≥1000/µL and platelets ≥100,000/µL. C1 extramedullary disease status was required. CRi was defined as CR except with ANC <1000/µL and/or platelets <100,000/µL.
Time Frame: From screening to progressive disease or another induction therapy started, up to approximately 2 years
Population: Safety analysis set
Measure: Number (90% Confidence Interval); unit: Percentage of Partcicipants
Arm/Group | Phase 2: IV Inotuzumab Ozogamicin 1.8mg/m^2
Number analyzed (Participants) | 35
Percentage of Partcicipants | 68.6 [53.39 to 81.27]

4. Primary Outcome: Percentage of Participants With CR, CRi or PR During the Phase 1 Expansion Phase
Description: CR was defined as a disappearance of leukemia as indicated by <5% marrow blasts and the absence of peripheral blood leukemic blasts, with recovery of hematopoiesis defined by ANC ≥1000/µL and platelets ≥100,000/µL. C1 extramedullary disease status was required. CRi was defined as CR except with ANC <1000/µL and/or platelets <100,000/µL. PR was defined as an improved or no worsening of acute lymphocytic leukemia as indicated by no peripheral blood blasts, and either or both of the following: at least a 50% decrease in the marrow blast percentage, compared to the pre-treatment value, and marrow blast percentage ≥5% and ≤25% and/or C2 extramedullary disease status.
Time Frame: From screening to progressive disease or another induction therapy started, up to approximately 2 years
Population: Safety analysis set
Measure: Number (95% Confidence Interval); unit: Percentage of Partcicipants
Arm/Group | Phase 1 - Expansion Phase: IV Inotuzumab Ozogamicin 1.8 mg/m^2
Number analyzed (Participants) | 13
Percentage of Partcicipants | 46.2 [19.22 to 74.87]

5. Secondary Outcome: Percentage of Participants With CR, CRi or PR in Phase 2
Description: as for outcome 4
Time Frame: From screening to progressive disease or another induction therapy started, up to approximately 2 years
Population: Safety analysis set
Measure: Number (95% Confidence Interval); unit: Percentage of Partcicipants
Arm/Group | Phase 2: IV Inotuzumab Ozogamicin 1.8mg/m^2
Number analyzed (Participants) | 35
Percentage of Partcicipants | 74.3 [56.74 to 87.51]

6. Secondary Outcome: Number of Participants With Minimal Residual Disease (MRD) Negativity in Participants Achieving CR and CRi
Description: MRD negativity was defined as <0.01% mononuclear cells.
Time Frame: From screening to progressive disease or another induction therapy started, up to approximately 2 years
Population: Number of participants who achieved CR and CRi
Measure: Number; unit: Participants
Arm/Group | Phase 1 - Dose-Finding: IV Inotuzumab Ozogamicin 1.2 mg/m^2 | Phase 1 - Dose Finding: IV Inotuzumab Ozogamicin 1.6 mg/m^2 | Phase 1 - Dose-Finding: IV Inotuzumab Ozogamicin 1.8 mg/m^2 | Phase 1 - Expansion Phase: IV Inotuzumab Ozogamicin 1.8 mg/m^2 | Phase 2: IV Inotuzumab Ozogamicin 1.8mg/m^2 | All Doses
Number analyzed (Participants) | 2 | 9 | 8 | 6 | 24 | 49
Participants | 2 | 8 | 8 | 5 | 18 | 41

7. Secondary Outcome: Percentage of Participants With CR or CRi by Cytogenetic Category
Description: as for outcome 3
Time Frame: From screening to progressive disease or another induction therapy started, up to approximately 2 years
Population: Safety analysis set (n refers to number of participants evaluated)
Measure: Number; unit: Percentage of Participants
Arm/Group | All Doses
Number analyzed (Participants) | 72
Percentage of Participants
  Normal (n=13) | 86.7
  Complex (n=10) | 66.7
  Ph+ (n=9) | 56.3
  Other (n=13) | 65.0
  Unknown (n=3) | 75.0
  Missing (n=1) | 50

8. Secondary Outcome: Percentage of Participants Who Had a Post-Treatment Stem-Cell Transplant (SCT)
Description: Post-treatment SCT rate was defined as the percentage of participants who underwent SCT following treatment with inotuzumab ozogamicin.
Time Frame: Up to approximately 2 years from first dose
Population: Safety analysis set
Measure: Number; unit: Percentage of Particicpants
Arm/Group | Phase 1 - Dose-Finding: IV Inotuzumab Ozogamicin 1.2 mg/m^2 | Phase 1 - Dose Finding: IV Inotuzumab Ozogamicin 1.6 mg/m^2 | Phase 1 - Dose-Finding: IV Inotuzumab Ozogamicin 1.8 mg/m^2 | Phase 1 - Expansion Phase: IV Inotuzumab Ozogamicin 1.8 mg/m^2 | Phase 2: IV Inotuzumab Ozogamicin 1.8mg/m^2 | All Doses
Number analyzed (Participants) | 3 | 12 | 9 | 13 | 35 | 72
Percentage of Particicpants | 0 | 75.0 | 44.4 | 23.1 | 22.9 | 33.3

9. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from Cycle 1 Day 1 to first documentation of PFS event (earliest date of objective progression [PD], treatment discontinuation due to global deterioration of health status, subsequent induction or transplant after best response of PR or resistant disease, relapse after CR or CRi, or death due to any cause). Participants last known to be 1) alive and 2) without a PFS event, were censored at the date of the last disease assessment that verified lack of event.
Time Frame: Up to approximately 2 years from first dose
Population: Safety analysis set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 1 - Dose-Finding: IV Inotuzumab Ozogamicin 1.2 mg/m^2 | Phase 1 - Dose Finding: IV Inotuzumab Ozogamicin 1.6 mg/m^2 | Phase 1 - Dose-Finding: IV Inotuzumab Ozogamicin 1.8 mg/m^2 | Phase 1 - Expansion Phase: IV Inotuzumab Ozogamicin 1.8 mg/m^2 | Phase 2: IV Inotuzumab Ozogamicin 1.8mg/m^2 | All Doses
Number analyzed (Participants) | 3 | 12 | 9 | 13 | 35 | 72
Months | 5.5 [2.1 to 6.4] | NA [1.4 to NA] — Median and upper 95% CI may not have been reached at the time of data analysis. | 8.8 [1.3 to 16.7] | 1.9 [1.0 to 5.0] | 3.7 [2.6 to 4.7] | 3.9 [3.0 to 5.4]

10. Secondary Outcome: Duration of Remission (DoR1) for Participants Who Achieved CR or CRi
Description: DoR1 was defined for participants who responded as the time from the date of first documentation of Complete Hematologic Response (CR or CRi) to the date of the first documentation of relapse after CR or CRi, treatment discontinuation due to global deterioration of health status) or to death due to any cause. Participants last known to be 1) alive and 2) without a DoR1 event, were censored at the date of the last disease assessment that verified lack of event.
Time Frame: Up to approximately 2 years from first dose
Population: All participants who achieved CR or CRi
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 1 - Dose-Finding: IV Inotuzumab Ozogamicin 1.2 mg/m^2 | Phase 1 - Dose Finding: IV Inotuzumab Ozogamicin 1.6 mg/m^2 | Phase 1 - Dose-Finding: IV Inotuzumab Ozogamicin 1.8 mg/m^2 | Phase 1 - Expansion Phase: IV Inotuzumab Ozogamicin 1.8 mg/m^2 | Phase 2: IV Inotuzumab Ozogamicin 1.8mg/m^2 | All Doses
Number analyzed (Participants) | 2 | 9 | 8 | 6 | 24 | 49
Months | 4.7 [4.6 to 4.8] | NA [0.7 to NA] — Median and upper 95% CI may not have been reached at the time of data analysis. | 10.8 [1.2 to NA] — Upper 95% CI may not have been reached at the time of data analysis. | 7.1 [2.1 to NA] — Upper 95% CI may not have been reached at the time of data analysis. | 3.8 [2.2 to 5.8] | 4.8 [3.8 to 7.0]

11. Secondary Outcome: Duration of Response (DoR) for Participants Who Achieved CR/CRi or PR
Description: DoR was defined for participants who respond as the time from the date of first documentation of Hematologic Response (CR, CRi, or PR) to the date of the first documentation of DoR event (earliest date of PD, treatment discontinuation due to global deterioration of health status, first induction therapy or transplant after PR, relapse after CR or CRi or death due to any cause). Participants last known to be 1) alive and 2) without a DoR event, were censored at the date of the last disease assessment that verified lack of event.
Time Frame: Up to approximately 2 years from first dose
Population: All participants who achieved CR, CRi or PR.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Phase 1 - Dose-Finding: IV Inotuzumab Ozogamicin 1.2 mg/m^2 | Phase 1 - Dose Finding: IV Inotuzumab Ozogamicin 1.6 mg/m^2 | Phase 1 - Dose-Finding: IV Inotuzumab Ozogamicin 1.8 mg/m^2 | Phase 1 - Expansion Phase: IV Inotuzumab Ozogamicin 1.8 mg/m^2 | Phase 2: IV Inotuzumab Ozogamicin 1.8mg/m^2 | All Doses
Number analyzed (Participants) | 2 | 11 | 8 | 6 | 26 | 53
Weeks | 20.50 [20.1 to 20.9] | NA [3.1 to NA] — Median and upper 95% CI may not have been reached at the time of data analysis. | 46.93 [7.6 to NA] — Upper 95% CI may not have been reached at the time of data analysis. | 31.07 [12.1 to NA] — Upper 95% CI may not have been reached at the time of data analysis. | 16.57 [9.9 to 24.0] | 18.71 [12.6 to 25.6]

12. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from Cycle 1 Day 1 to date of death due to any cause. If death was not documented, censoring occurred at the date at which the participant was last known to be alive.
Time Frame: Up to approximately 2 years from first dose
Population: Safety analysis set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 1 - Dose-Finding: IV Inotuzumab Ozogamicin 1.2 mg/m^2 | Phase 1 - Dose Finding: IV Inotuzumab Ozogamicin 1.6 mg/m^2 | Phase 1 - Dose-Finding: IV Inotuzumab Ozogamicin 1.8 mg/m^2 | Phase 1 - Expansion Phase: IV Inotuzumab Ozogamicin 1.8 mg/m^2 | Phase 2: IV Inotuzumab Ozogamicin 1.8mg/m^2 | All Doses
Number analyzed (Participants) | 3 | 12 | 9 | 13 | 35 | 72
Months | 9.2 [2.1 to 11.3] | NA [2.6 to NA] — Median and upper 95% CI may not have been reached at the time of data analysis. | 16.5 [2.6 to NA] — Upper 95% CI may not have been reached at the time of data analysis. | 5.8 [3.5 to 10.8] | 6.4 [4.5 to 7.9] | 7.4 [5.7 to 9.2]

13. Secondary Outcome: Time to Remission for Participants Who Achieved CR or CRi
Description: Time to remission was defined as the time from the date of first dose of study drug to the date of first documentation of hematologic remission (CR or CRi) in participants achieving remission during study therapy.
Time Frame: Up to approximately 2 years from first dose
Population: All participants who achieved CR or CRi
Measure: Median (Full Range); unit: Days
Arm/Group | Phase 1 - Dose-Finding: IV Inotuzumab Ozogamicin 1.2 mg/m^2 | Phase 1 - Dose Finding: IV Inotuzumab Ozogamicin 1.6 mg/m^2 | Phase 1 - Dose-Finding: IV Inotuzumab Ozogamicin 1.8 mg/m^2 | Phase 1 - Expansion Phase: IV Inotuzumab Ozogamicin 1.8 mg/m^2 | Phase 2: IV Inotuzumab Ozogamicin 1.8mg/m^2 | All Doses
Number analyzed (Participants) | 2 | 9 | 8 | 6 | 24 | 49
Days | 39.0 (24.04) [22 to 56] | 29.0 (12.60) [22 to 59] | 38.0 (19.88) [22 to 78] | 27.0 (29.18) [21 to 85] | 25.5 (22.12) [15 to 91] | 27.0 (20.75) [15 to 91]

14. Secondary Outcome: Time to Response for Participants Who Achieved CR/CRi or PR
Description: Time to response was defined as the time from the date of first dose of study drug to the date of first documentation of hematologic response (CR, CRi, or PR).
Time Frame: Up to approximately 2 years from first dose
Population: All participants who achieved CR, CRi or PR.
Measure: Median (Full Range); unit: Days
Arm/Group | Phase 1 - Dose-Finding: IV Inotuzumab Ozogamicin 1.2 mg/m^2 | Phase 1 - Dose Finding: IV Inotuzumab Ozogamicin 1.6 mg/m^2 | Phase 1 - Dose-Finding: IV Inotuzumab Ozogamicin 1.8 mg/m^2 | Phase 1 - Expansion Phase: IV Inotuzumab Ozogamicin 1.8 mg/m^2 | Phase 2: IV Inotuzumab Ozogamicin 1.8mg/m^2 | All Doses
Number analyzed (Participants) | 2 | 11 | 8 | 6 | 26 | 53
Days | 39.0 (24.04) [22 to 56] | 29.0 (9.01) [22 to 49] | 27.0 (20.66) [20 to 78] | 24.0 (10.09) [21 to 48] | 23.0 (10.22) [15 to 58] | 25.0 (12.45) [15 to 78]

15. Secondary Outcome: Time to MRD Negativity for Participants Who Achieved CR or CRi
Description: Time to MRD negativity was defined as the time from the date of first dose of study drug to the date of first documentation of MRD negativity.
Time Frame: Screening, Day 21 of Cycles 1 to 6 and up to 4 to 6 weeks after the last dose (up to 34 weeks)
Population: All participants who achieved CR/CRi and MRD negativity.
Measure: Median (Full Range); unit: Days
Arm/Group | Phase 1 - Dose-Finding: IV Inotuzumab Ozogamicin 1.2 mg/m^2 | Phase 1 - Dose Finding: IV Inotuzumab Ozogamicin 1.6 mg/m^2 | Phase 1 - Dose-Finding: IV Inotuzumab Ozogamicin 1.8 mg/m^2 | Phase 1 - Expansion Phase: IV Inotuzumab Ozogamicin 1.8 mg/m^2 | Phase 2: IV Inotuzumab Ozogamicin 1.8mg/m^2 | All Doses
Number analyzed (Participants) | 2 | 8 | 8 | 5 | 18 | 41
Days | 98.5 (0.71) [98 to 99] | 32.0 (15.17) [22 to 64] | 30.0 (50.54) [22 to 141] | 25.0 (48.09) [21 to 134] | 25.5 (18.66) [21 to 80] | 29.0 (32.73) [21 to 141]

16. Secondary Outcome: Duration of Follow-Up
Description: Duration of follow-up was defined as the time from the date of first dose of study drug to the date of last contact for participants known to be alive.
Time Frame: From first dose up to approximately 2 years
Population: Participants who were alive
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 1 - Dose-Finding: IV Inotuzumab Ozogamicin 1.2 mg/m^2 | Phase 1 - Dose Finding: IV Inotuzumab Ozogamicin 1.6 mg/m^2 | Phase 1 - Dose-Finding: IV Inotuzumab Ozogamicin 1.8 mg/m^2 | Phase 1 - Expansion Phase: IV Inotuzumab Ozogamicin 1.8 mg/m^2 | Phase 2: IV Inotuzumab Ozogamicin 1.8mg/m^2 | All Doses
Number analyzed (Participants) | 0 | 6 | 3 | 3 | 5 | 17
Months |  | 24.0 [22.9 to 29.7] | 25.7 [24.1 to 26.5] | 24.1 [23.9 to 26.9] | 24.2 [6.8 to 24.5] | 24.1 [24.0 to 24.5]

17. Secondary Outcome: Percentage of Cluster of Differentiation-22 Positive (CD22+) Leukemic Blasts in Abnormal B Cells in Blood by Visit
Description: CD22+ leukemic blasts assessed in abnormal B cells from blood (data from central laboratories only).
Time Frame: Pre-dose on Days 1 and 15 of Cycles 1 and 2, and Day 1 of Cycle 4
Population: Safety analysis set
Measure: Median (Full Range); unit: Percentage of CD22+
Arm/Group | Phase 1 - Dose-Finding: IV Inotuzumab Ozogamicin 1.2 mg/m^2 | Phase 1 - Dose Finding: IV Inotuzumab Ozogamicin 1.6 mg/m^2 | Phase 1 - Dose-Finding: IV Inotuzumab Ozogamicin 1.8 mg/m^2 | Phase 1 - Expansion Phase: IV Inotuzumab Ozogamicin 1.8 mg/m^2 | Phase 2: IV Inotuzumab Ozogamicin 1.8mg/m^2 | All Doses
Number analyzed (Participants) | 3 | 12 | 9 | 13 | 35 | 72
Percentage of CD22+
  Screening | NA [NA to NA] — Median and CI not determined since n = 0 | NA [NA to NA] — Median and CI not determined since n = 0 | NA [NA to NA] — Median and CI not determined since n = 0 | 93.7 [88 to 100] | NA [NA to NA] — Median and CI not determined since n = 0 | 93.7 [88 to 100]
  Cycle 1 Day 1 | 99.7 [57 to 100] | 98.1 [67 to 100] | 98.4 [0 to 100] | 96.4 [65 to 100] | 98.7 [0 to 100] | 98.0 [0 to 100]
  Cycle 1 Day 15 | 66.2 [31 to 99] | 79.0 [0 to 100] | 0.0 [0 to 99] | 71.4 [0 to 100] | 74.8 [0 to 100] | 69.9 [0 to 100]
  Cycle 2 Day 1 | 52.0 [6 to 100] | 0.0 [0 to 100] | 0.0 [0 to 92] | 2.8 [0 to 100] | 0.0 [0 to 100] | 0.0 [0 to 100]
  Cycle 2 Day 15 | 0.0 [0 to 0] | 0.0 [0 to 98] | 0.0 [0 to 0] | 0.5 [0 to 99] | 0.0 [0 to 100] | 0.0 [0 to 100]
  Cycle 4 Day 1 | 49.2 [0 to 100] | 0.0 [0 to 0] | 0.0 [0 to 73] | 0.0 [0 to 38] | 0.0 [0 to 100] | 0.0 [0 to 100]
  End of Treatment | 99.0 [99 to 99] | NA [NA to NA] — Median and CI not determined since n = 0 | NA [NA to NA] — Median and CI not determined since n = 0 | NA [NA to NA] — Median and CI not determined since n = 0 | NA [NA to NA] — Median and CI not determined since n = 0 | 99.0 [99 to 99]

18. Secondary Outcome: Percentage of CD22+ Leukemic Blasts in Abnormal B Cells in Bone Marrow by Visit
Description: CD22+ leukemic blasts assessed in abnormal B cells from bone marrow (data from central laboratories only).
Time Frame: Pre-dose on Days 1 and 15 of Cycles 1 and 2, and Day 1 of Cycle 4
Population: Safety analysis set
Measure: Median (Full Range); unit: Percentage of CD22+
Arm/Group | Phase 1 - Dose-Finding: IV Inotuzumab Ozogamicin 1.2 mg/m^2 | Phase 1 - Dose Finding: IV Inotuzumab Ozogamicin 1.6 mg/m^2 | Phase 1 - Dose-Finding: IV Inotuzumab Ozogamicin 1.8 mg/m^2 | Phase 1 - Expansion Phase: IV Inotuzumab Ozogamicin 1.8 mg/m^2 | Phase 2: IV Inotuzumab Ozogamicin 1.8mg/m^2 | All Doses
Number analyzed (Participants) | 3 | 12 | 9 | 13 | 35 | 72
Percentage of CD22+
  Screening | 99.6 [96 to 100] | 98.7 [31 to 100] | 98.4 [97 to 100] | 95.1 [52 to 100] | 99.2 [78 to 100] | 99.0 [31 to 100]
  Cycle 1 Day 21 | NA [NA to NA] — Median and CI not determined since n = 0 | NA [NA to NA] — Median and CI not determined since n = 0 | 99 [99 to 99] | 56.5 [39 to 74] | 70.7 [0 to 100] | 72.3 [0 to 100]
  Cycle 1 Day 28 | 75.5 [52 to 99] | 54.1 [0 to 100] | 26.5 [0 to 99] | 74.1 [0 to 100] | 94.5 [20 to 100] | 56.6 [0 to 100]
  Cycle 2 Day 21 | NA [NA to NA] — Median and CI not determined since n = 0 | 0.0 [0 to 0] | NA [NA to NA] — Median and CI not determined since n = 0 | NA [NA to NA] — Median and CI not determined since n = 0 | 0.0 [0 to 96] | 0.0 [0 to 96]
  Cycle 2 Day 28 | 52.9 [6 to 100] | 0.0 [0 to 31] | 0.0 [0 to 72] | 2.9 [0 to 100] | 6.8 [0 to 78] | 0.0 [0 to 100]
  Cycle 3 Day 21 | NA [NA to NA] — Median and CI not determined since n = 0 | NA [NA to NA] — Median and CI not determined since n = 0 | 0.0 [0 to 0] | 0.0 [0 to 0] | 0.0 [0 to 71] | 0.0 [0 to 71]
  Cycle 3 Day 28 | 50.0 [0 to 100] | 0.0 [0 to 0] | 0.0 [0 to 13] | 0.0 [0 to 78] | 25.1 [0 to 50] | 0.0 [0 to 100]
  Cycle 4 Day 21 | 97 [97 to 97] | NA [NA to NA] — Median and CI not determined since n = 0 | NA [NA to NA] — Median and CI not determined since n = 0 | NA [NA to NA] — Median and CI not determined since n = 0 | 11.6 [0 to 45] | 23.2 [0 to 97]
  Cycle 4 Day 28 | 0.0 [0 to 0] | 0.0 [0 to 0] | 14.3 [2 to 27] | 29.4 [0 to 59] | 36 [36 to 36] | 1.9 [0 to 59]
  Cycle 5 Day 21 | NA [NA to NA] — Median and CI not determined since n = 0 | NA [NA to NA] — Median and CI not determined since n = 0 | NA [NA to NA] — Median and CI not determined since n = 0 | 0.0 [0 to 0] | 66.4 [48 to 85] | 48.1 [0 to 85]
  Cycle 5 Day 28 | 0.0 [0 to 0] | NA [NA to NA] — Median and CI not determined since n = 0 | NA [NA to NA] — Median and CI not determined since n = 0 | 79.1 [0 to 99] | NA [NA to NA] — Median and CI not determined since n = 0 | 39.6 [0 to 99]
  Cycle 6 Day 21 | NA [NA to NA] — Median and CI not determined since n = 0 | NA [NA to NA] — Median and CI not determined since n = 0 | NA [NA to NA] — Median and CI not determined since n = 0 | 0.0 [0 to 0] | 74 [74 to 74] | 0.0 [0 to 74]
  End of Treatment | 100 [100 to 100] | 0.0 [0 to 4] | 0.0 [0 to 0] | 6.6 [2 to 11] | 0.0 [0 to 94] | 0.0 [0 to 100]

19. Secondary Outcome: Messenger Ribonucleic Acid (mRNA) Gene Expression
Description: Optional blood samples for pharmacogenomic parameters were collected during Cycle 1 prior to the start of the inotuzumab ozogamicin infusion (0 hours) and 1 hour post-dose (original Final Protocol and Protocol Amendments 1 and 2) or 3 hours post-dose (Protocol Amendments 3 and 4) on Day 1 and Day 15 from those participants who provided consent. Gene expression analysis of samples collected pre- and post-dosing was performed using 96-gene TaqMan® low density array cards to examine the concordance between clinical outcome and expression of genes such as those involved in DNA damage response, apoptosis, B-cell antigen expression, glutathione metabolism, drug transport and the phosphoinositide 3-kinase/mammalian target of rapamycin pathway. Expression for each gene was reported as a normalized value, 2^-change in (∆) threshold cycle (Ct), where ∆Ct is Ct^target gene minus Ct^reference genes, averaged.
Time Frame: Predose and postdose on Days 1 and 15 of Cycle 1
Population: Pharmacogenomics population - included all enrolled participants who received at least 1 dose of any study drug, and had at least 1 biomarker parameter from the corresponding assay sample with both a baseline and post-treatment assessment.
Measure: Median (Full Range); unit: Fold expression
Groups:
- Pharmacogenomics Population: All participants who gave consent for the optional blood sample for pharmacogenomic analyses, received at least 1 dose of any study drug, and had at least 1 biomarker parameter from the corresponding assay sample with both a baseline and post-treatment assessment.
Arm/Group | Pharmacogenomics Population
Number analyzed (Participants) | 55
Fold expression
  ABCB1: Cycle 1 Day 1, Baseline (n=55) | 0.00421 [0.0002 to 0.0217]
  ABCB1: Cycle 1 Day 1, Post-dose (n=51) | 0.00440 [0.0003 to 0.0313]
  ABCB1: Cycle 1 Day 15, 0 hours (n=48) | 0.00746 [0.0004 to 0.0218]
  ABCB1: Cycle 1 Day 15, Post-dose (n=46) | 0.00783 [0.0005 to 0.0364]
  ABCC1: Cycle 1 Day 1, Baseline (n=55) | 0.01983 [0.0041 to 0.0885]
  ABCC1: Cycle 1 Day 1, Post-dose (n=52) | 0.02245 [0.0044 to 0.0737]
  ABCC1: Cycle 1 Day 15, 0 hours (n=48) | 0.01453 [0.0062 to 0.0413]
  ABCC1: Cycle 1 Day 15, Post-dose (n=46) | 0.01497 [0.0042 to 0.0578]
  ABCC2: Cycle 1 Day 1, Baseline (n=53) | 0.00064 [0.0002 to 0.0020]
  ABCC2: Cycle 1 Day 1, Post-dose (n=48) | 0.00072 [0.0002 to 0.0020]
  ABCC2: Cycle 1 Day 15, 0 hours (n=40) | 0.00072 [0.0002 to 0.0015]
  ABCC2: Cycle 1 Day 15, Post-dose (n=38) | 0.00078 [0.0003 to 0.0023]
  ABCG2: Cycle 1 Day 1, Baseline (n=55) | 0.00491 [0.0003 to 0.0509]
  ABCG2: Cycle 1 Day 1, Post-dose (n=51) | 0.00660 [0.0002 to 0.0431]
  ABCG2: Cycle 1 Day 15, 0 hours (n=46) | 0.01582 [0.0014 to 0.0818]
  ABCG2: Cycle 1 Day 15, Post-dose (n=45) | 0.01845 [0.0010 to 0.0921]
  ABL1: Cycle 1 Day 1, Baseline (n=55) | 0.03297 [0.0027 to 0.1982]
  ABL1: Cycle 1 Day 1, Post-dose (n=52) | 0.02899 [0.0032 to 0.1382]
  ABL1: Cycle 1 Day 15, 0 hours (n=48) | 0.01369 [0.0043 to 0.0632]
  ABL1: Cycle 1 Day 15, Post-dose (n=46) | 0.01381 [0.0032 to 0.0783]
  ABL2: Cycle 1 Day 1, Baseline (n=55) | 0.00916 [0.0029 to 0.0329]
  ABL2: Cycle 1 Day 1, Post-dose (n=52) | 0.00867 [0.0021 to 0.0268]
  ABL2: Cycle 1 Day 15, 0 hours (n=48) | 0.00613 [0.0032 to 0.0184]
  ABL2: Cycle 1 Day 15, Post-dose (n=46) | 0.00547 [0.0029 to 0.0224]
  ACTB: Cycle 1 Day 1, Baseline (n=55) | 1.73899 [0.5853 to 4.0764]
  ACTB: Cycle 1 Day 1, Post-dose (n=52) | 1.95092 [0.7314 to 3.3585]
  ACTB: Cycle 1 Day 15, 0 hours (n=48) | 2.14694 [1.3915 to 5.3955]
  ACTB: Cycle 1 Day 15, Post-dose (n=46) | 2.11584 [1.3279 to 7.3316]
  AKT1: Cycle 1 Day 1, Baseline (n=55) | 0.03212 [0.0112 to 0.0793]
  AKT1: Cycle 1 Day 1, Post-dose (n=52) | 0.03164 [0.0116 to 0.0738]
  AKT1: Cycle 1 Day 15, 0 hours (n=48) | 0.02740 [0.0108 to 0.0572]
  AKT1: Cycle 1 Day 15, Post-dose (n=46) | 0.02987 [0.0078 to 0.0672]
  ALG5: Cycle 1 Day 1, Baseline (n=55) | 0.00455 [0.0004 to 0.0206]
  ALG5: Cycle 1 Day 1, Post-dose (n=52) | 0.00419 [0.0007 to 0.0173]
  ALG5: Cycle 1 Day 15, 0 hours (n=48) | 0.00302 [0.0013 to 0.0064]
  ALG5: Cycle 1 Day 15, Post-dose (n=46) | 0.00265 [0.0006 to 0.0060]
  APAF1: Cycle 1 Day 1, Baseline (n=55) | 0.03880 [0.0074 to 0.0896]
  APAF1: Cycle 1 Day 1, Post-dose (n=52) | 0.03740 [0.0072 to 0.1051]
  APAF1: Cycle 1 Day 15, 0 hours (n=48) | 0.03754 [0.0138 to 0.0763]
  APAF1: Cycle 1 Day 15, Post-dose (n=46) | 0.03708 [0.0128 to 0.0918]
  ATM: Cycle 1 Day 1, Baseline (n=55) | 0.06441 [0.0121 to 0.1845]
  ATM: Cycle 1 Day 1, Post-dose (n=52) | 0.06615 [0.0125 to 0.1497]
  ATM: Cycle 1 Day 15, 0 hours (n=48) | 0.06927 [0.0297 to 0.1439]
  ATM: Cycle 1 Day 15, Post-dose (n=46) | 0.05951 [0.0262 to 0.1247]
  ATRX: Cycle 1 Day 1, Baseline (n=55) | 0.06123 [0.0177 to 0.2406]
  ATRX: Cycle 1 Day 1, Post-dose (n=52) | 0.05679 [0.0194 to 0.2183]
  ATRX: Cycle 1 Day 15, 0 hours (n=48) | 0.05456 [0.0179 to 0.1074]
  ATRX: Cycle 1 Day 15, Post-dose (n=46) | 0.05662 [0.0211 to 0.1142]
  B2M: Cycle 1 Day 1, Baseline (n=55) | 3.81650 [1.2559 to 9.9074]
  B2M: Cycle 1 Day 1, Post-dose (n=52) | 3.89919 [1.2108 to 11.9448]
  B2M: Cycle 1 Day 15, 0 hours (n=48) | 5.97465 [1.1943 to 10.8448]
  B2M: Cycle 1 Day 15, Post-dose (n=46) | 6.21338 [1.5174 to 12.9707]
  BAD: Cycle 1 Day 1, Baseline (n=55) | 0.00099 [0.0004 to 0.0053]
  BAD: Cycle 1 Day 1, Post-dose (n=52) | 0.00100 [0.0003 to 0.0067]
  BAD: Cycle 1 Day 15, 0 hours (n=47) | 0.00085 [0.0003 to 0.0021]
  BAD: Cycle 1 Day 15, Post-dose (n=43) | 0.00077 [0.0004 to 0.0026]
  BAK1: Cycle 1 Day 1, Baseline (n=55) | 0.01991 [0.0031 to 0.2253]
  BAK1: Cycle 1 Day 1, Post-dose (n=52) | 0.01658 [0.0024 to 0.1570]
  BAK1: Cycle 1 Day 15, 0 hours (n=48) | 0.01490 [0.0050 to 0.0313]
  BAK1: Cycle 1 Day 15, Post-dose (n=46) | 0.01405 [0.0045 to 0.0302]
  BAX: Cycle 1 Day 1, Baseline (n=55) | 0.07686 [0.0290 to 0.1825]
  BAX: Cycle 1 Day 1, Post-dose (n=52) | 0.07420 [0.0284 to 0.1904]
  BAX: Cycle 1 Day 15, 0 hours (n=48) | 0.07107 [0.0346 to 0.1387]
  BAX: Cycle 1 Day 15, Post-dose (n=46) | 0.06543 [0.0304 to 0.1316]
  BBC3: Cycle 1 Day 1, Baseline (n=55) | 0.01174 [0.0031 to 0.0445]
  BBC3: Cycle 1 Day 1, Post-dose (n=52) | 0.01197 [0.0044 to 0.0384]
  BBC3: Cycle 1 Day 15, 0 hours (n=48) | 0.01470 [0.0052 to 0.0335]
  BBC3: Cycle 1 Day 15, Post-dose (n=46) | 0.01449 [0.0061 to 0.0390]
  BCL2: Cycle 1 Day 1, Baseline (n=55) | 0.02425 [0.0021 to 0.0958]
  BCL2: Cycle 1 Day 1, Post-dose (n=52) | 0.02200 [0.0024 to 0.1014]
  BCL2: Cycle 1 Day 15, 0 hours (n=48) | 0.01979 [0.0037 to 0.0703]
  BCL2: Cycle 1 Day 15, Post-dose (n=46) | 0.01648 [0.0042 to 0.0851]
  BCL2L1: Cycle 1 Day 1, Baseline (n=55) | 0.83473 [0.0227 to 11.2775]
  BCL2L1: Cycle 1 Day 1, Post-dose (n=52) | 1.12931 [0.0200 to 14.5203]
  BCL2L1: Cycle 1 Day 15, 0 hours (n=48) | 3.05721 [0.0236 to 15.0024]
  BCL2L1: Cycle 1 Day 15, Post-dose (n=46) | 3.98955 [0.0220 to 18.3879]
  BCL2L11: Cycle 1 Day 1, Baseline (n=55) | 0.03003 [0.0025 to 0.1197]
  BCL2L11: Cycle 1 Day 1, Post-dose (n=52) | 0.02970 [0.0029 to 0.0916]
  BCL2L11: Cycle 1 Day 15, 0 hours (n=48) | 0.03865 [0.0151 to 0.0817]
  BCL2L11: Cycle 1 Day 15, Post-dose (n=46) | 0.04259 [0.0164 to 0.0825]
  BCR: Cycle 1 Day 1, Baseline (n=7) | 0.02294 [0.0006 to 0.0858]
  BCR: Cycle 1 Day 1, Post-dose (n=5) | 0.02135 [0.0008 to 0.0967]
  BCR: Cycle 1 Day 15, 0 hours (n=3) | 0.00116 [0.0003 to 0.0108]
  BCR: Cycle 1 Day 15, Post-dose (n=2) | 0.00817 [0.0013 to 0.0150]
  BID: Cycle 1 Day 1, Baseline (n=55) | 0.01794 [0.0076 to 0.0458]
  BID: Cycle 1 Day 1, Post-dose (n=52) | 0.01528 [0.0060 to 0.0436]
  BID: Cycle 1 Day 15, 0 hours (n=48) | 0.01619 [0.0071 to 0.0313]
  BID: Cycle 1 Day 15, Post-dose (n=46) | 0.01448 [0.0043 to 0.0518]
  BIK: Cycle 1 Day 1, Baseline (n=52) | 0.00137 [0.0001 to 0.0220]
  BIK: Cycle 1 Day 1, Post-dose (n=49) | 0.00143 [0.0001 to 0.0228]
  BIK: Cycle 1 Day 15, 0 hours (n=42) | 0.00093 [0.0005 to 0.0038]
  BIK: Cycle 1 Day 15, Post-dose (n=39) | 0.00095 [0.0004 to 0.0049]
  BMF: Cycle 1 Day 1, Baseline (n=55) | 0.00604 [0.0011 to 0.0579]
  BMF: Cycle 1 Day 1, Post-dose (n=52) | 0.00705 [0.0009 to 0.0807]
  BMF: Cycle 1 Day 15, 0 hours (n=47) | 0.00333 [0.0010 to 0.0156]
  BMF: Cycle 1 Day 15, Post-dose (n=46) | 0.00341 [0.0006 to 0.0429]
  BRCA1: Cycle 1 Day 1, Baseline (n=55) | 0.00628 [0.0017 to 0.0395]
  BRCA1: Cycle 1 Day 1, Post-dose (n=52) | 0.00691 [0.0019 to 0.0367]
  BRCA1: Cycle 1 Day 15, 0 hours (n=48) | 0.00385 [0.0019 to 0.0133]
  BRCA1: Cycle 1 Day 15, Post-dose (n=46) | 0.00416 [0.0024 to 0.0175]
  BRCA2: Cycle 1 Day 1, Baseline (n=50) | 0.00059 [0.0002 to 0.0023]
  BRCA2: Cycle 1 Day 1, Post-dose (n=44) | 0.00067 [0.0002 to 0.0020]
  BRCA2: Cycle 1 Day 15, 0 hours (n=34) | 0.00045 [0.0003 to 0.0015]
  BRCA2: Cycle 1 Day 15, Post-dose (n=35) | 0.00049 [0.0003 to 0.0012]
  CA6: Cycle 1 Day 1, Baseline (n=48) | 0.00104 [0.0001 to 0.1076]
  CA6: Cycle 1 Day 1, Post-dose (n=42) | 0.00196 [0.0000 to 0.1364]
  CA6: Cycle 1 Day 15, 0 hours (n=35) | 0.00130 [0.0002 to 0.0425]
  CA6: Cycle 1 Day 15, Post-dose (n=34) | 0.00119 [0.0003 to 0.0576]
  CASP2: Cycle 1 Day 1, Baseline (n=55) | 0.04235 [0.0161 to 0.1661]
  CASP2: Cycle 1 Day 1, Post-dose (n=52) | 0.04162 [0.0141 to 0.1175]
  CASP2: Cycle 1 Day 15, 0 hours (n=48) | 0.03287 [0.0201 to 0.1092]
  CASP2: Cycle 1 Day 15, Post-dose (n=46) | 0.03283 [0.0190 to 0.1097]
  CASP3: Cycle 1 Day 1, Baseline (n=55) | 0.02380 [0.0091 to 0.0608]
  CASP3: Cycle 1 Day 1, Post-dose (n=52) | 0.02353 [0.0046 to 0.0741]
  CASP3: Cycle 1 Day 15, 0 hours (n=48) | 0.02168 [0.0102 to 0.0404]
  CASP3: Cycle 1 Day 15, Post-dose (n=46) | 0.02030 [0.0068 to 0.0429]
  CASP7: Cycle 1 Day 1, Baseline (n=55) | 0.01271 [0.0032 to 0.0364]
  CASP7: Cycle 1 Day 1, Post-dose (n=52) | 0.01354 [0.0024 to 0.0278]
  CASP7: Cycle 1 Day 15, 0 hours (n=48) | 0.00923 [0.0026 to 0.0235]
  CASP7: Cycle 1 Day 15, Post-dose (n=46) | 0.00833 [0.0016 to 0.0196]
  CASP9: Cycle 1 Day 1, Baseline (n=55) | 0.00772 [0.0039 to 0.0211]
  CASP9: Cycle 1 Day 1, Post-dose (n=52) | 0.00732 [0.0033 to 0.0218]
  CASP9: Cycle 1 Day 15, 0 hours (n=48) | 0.00707 [0.0042 to 0.0120]
  CASP9: Cycle 1 Day 15, Post-dose (n=46) | 0.00715 [0.0037 to 0.0135]
  CCND1: Cycle 1 Day 1, Baseline (n=52) | 0.00091 [0.0001 to 0.0309]
  CCND1: Cycle 1 Day 1, Post-dose (n=49) | 0.00071 [0.0001 to 0.0153]
  CCND1: Cycle 1 Day 15, 0 hours (n=43) | 0.00080 [0.0002 to 0.0067]
  CCND1: Cycle 1 Day 15, Post-dose (n=37) | 0.00078 [0.0002 to 0.0044]
  CCNE1: Cycle 1 Day 1, Baseline (n=53) | 0.00311 [0.0003 to 0.0371]
  CCNE1: Cycle 1 Day 1, Post-dose (n=50) | 0.00331 [0.0005 to 0.0318]
  CCNE1: Cycle 1 Day 15, 0 hours (n=46) | 0.00234 [0.0004 to 0.0136]
  CCNE1: Cycle 1 Day 15, Post-dose (n=43) | 0.00217 [0.0002 to 0.0080]
  CD22: Cycle 1 Day 1, Baseline (n=55) | 0.04313 [0.0005 to 0.7239]
  CD22: Cycle 1 Day 1, Post-dose (n=51) | 0.03359 [0.0007 to 0.6010]
  CD22: Cycle 1 Day 15, 0 hours (n=35) | 0.00120 [0.0002 to 0.0559]
  CD22: Cycle 1 Day 15, Post-dose (n=32) | 0.00130 [0.0002 to 0.0684]
  CD24: Cycle 1 Day 1, Baseline (n=55) | 0.31881 [0.0232 to 2.6309]
  CD24: Cycle 1 Day 1, Post-dose (n=52) | 0.36597 [0.0237 to 3.0720]
  CD24: Cycle 1 Day 15, 0 hours (n=48) | 0.02968 [0.0019 to 0.5446]
  CD24: Cycle 1 Day 15, Post-dose (n=46) | 0.05363 [0.0036 to 0.6901]
  CD44: Cycle 1 Day 1, Baseline (n=55) | 0.25285 [0.1254 to 0.8904]
  CD44: Cycle 1 Day 1, Post-dose (n=52) | 0.23497 [0.0996 to 0.7828]
  CD44: Cycle 1 Day 15, 0 hours (n=48) | 0.27359 [0.1607 to 0.6984]
  CD44: Cycle 1 Day 15, Post-dose (n=46) | 0.22892 [0.1309 to 0.6394]
  CD70: Cycle 1 Day 1, Baseline (n=52) | 0.00194 [0.0000 to 0.0282]
  CD70: Cycle 1 Day 1, Post-dose (n=47) | 0.00170 [0.0001 to 0.0291]
  CD70: Cycle 1 Day 15, 0 hours (n=42) | 0.00225 [0.0002 to 0.0115]
  CD70: Cycle 1 Day 15, Post-dose (n=38) | 0.00169 [0.0001 to 0.0135]
  CDC25A: Cycle 1 Day 1, Baseline (n=53) | 0.00337 [0.0003 to 0.0290]
  CDC25A: Cycle 1 Day 1, Post-dose (n=50) | 0.00334 [0.0003 to 0.0292]
  CDC25A: Cycle 1 Day 15, 0 hours (n=45) | 0.00115 [0.0002 to 0.0100]
  CDC25A: Cycle 1 Day 15, Post-dose (n=36) | 0.00116 [0.0002 to 0.0098]
  CDK2: Cycle 1 Day 1, Baseline (n=55) | 0.02026 [0.0028 to 0.0786]
  CDK2: Cycle 1 Day 1, Post-dose (n=52) | 0.01883 [0.0031 to 0.0786]
  CDK2: Cycle 1 Day 15, 0 hours (n=48) | 0.01109 [0.0043 to 0.0389]
  CDK2: Cycle 1 Day 15, Post-dose (n=46) | 0.01118 [0.0039 to 0.0458]
  CDKN2A: Cycle 1 Day 1, Baseline (n=55) | 0.00675 [0.0002 to 0.7546]
  CDKN2A: Cycle 1 Day 1, Post-dose (n=52) | 0.00667 [0.0002 to 0.7308]
  CDKN2A: Cycle 1 Day 15, 0 hours (n=48) | 0.00676 [0.0001 to 0.0892]
  CDKN2A: Cycle 1 Day 15, Post-dose (n=46) | 0.00661 [0.0001 to 0.1001]
  CHEK2: Cycle 1 Day 1, Baseline (n=55) | 0.00257 [0.0008 to 0.0067]
  CHEK2: Cycle 1 Day 1, Post-dose (n=51) | 0.00224 [0.0008 to 0.0069]
  CHEK2: Cycle 1 Day 15, 0 hours (n=47) | 0.00206 [0.0006 to 0.0077]
  CHEK2: Cycle 1 Day 15, Post-dose (n=46) | 0.00234 [0.0009 to 0.0093]
  DAPK1: Cycle 1 Day 1, Baseline (n=55) | 0.02015 [0.0005 to 0.2850]
  DAPK1: Cycle 1 Day 1, Post-dose (n=52) | 0.02089 [0.0002 to 0.2330]
  DAPK1: Cycle 1 Day 15, 0 hours (n=48) | 0.01627 [0.0017 to 0.0447]
  DAPK1: Cycle 1 Day 15, Post-dose (n=46) | 0.01769 [0.0018 to 0.0544]
  DCLRE1C: Cycle 1 Day 1, Baseline (n=55) | 0.01404 [0.0030 to 0.0550]
  DCLRE1C: Cycle 1 Day 1, Post-dose (n=52) | 0.01226 [0.0028 to 0.0539]
  DCLRE1C: Cycle 1 Day 15, 0 hours (n=48) | 0.00845 [0.0034 to 0.0162]
  DCLRE1C: Cycle 1 Day 15, Post-dose (n=46) | 0.00875 [0.0031 to 0.0243]
  DDIT4L: Cycle 1 Day 1, Baseline (n=46) | 0.00091 [0.0001 to 0.0322]
  DDIT4L: Cycle 1 Day 1, Post-dose (n=41) | 0.00081 [0.0001 to 0.0169]
  DDIT4L: Cycle 1 Day 15, 0 hours (n=18) | 0.00058 [0.0002 to 0.0093]
  DDIT4L: Cycle 1 Day 15, Post-dose (n=13) | 0.00052 [0.0002 to 0.0115]
  EBF1: Cycle 1 Day 1, Baseline (n=55) | 0.02830 [0.0005 to 0.3909]
  EBF1: Cycle 1 Day 1, Post-dose (n=51) | 0.02492 [0.0006 to 0.3346]
  EBF1: Cycle 1 Day 15, 0 hours (n=35) | 0.00112 [0.0001 to 0.0761]
  EBF1: Cycle 1 Day 15, Post-dose (n=34) | 0.00112 [0.0002 to 0.1217]
  EEF1D: Cycle 1 Day 1, Baseline (n=55) | 0.00250 [0.0006 to 0.0115]
  EEF1D: Cycle 1 Day 1, Post-dose (n=52) | 0.00246 [0.0008 to 0.0108]
  EEF1D: Cycle 1 Day 15, 0 hours (n=48) | 0.00181 [0.0007 to 0.0051]
  EEF1D: Cycle 1 Day 15, Post-dose (n=46) | 0.00186 [0.0010 to 0.0059]
  FADD: Cycle 1 Day 1, Baseline (n=55) | 0.00436 [0.0022 to 0.0192]
  FADD: Cycle 1 Day 1, Post-dose (n=52) | 0.00487 [0.0018 to 0.0309]
  FADD: Cycle 1 Day 15, 0 hours (n=48) | 0.00434 [0.0022 to 0.0117]
  FADD: Cycle 1 Day 15, Post-dose (n=46) | 0.00477 [0.0024 to 0.0127]
  FAS: Cycle 1 Day 1, Baseline (n=55) | 0.02458 [0.0041 to 0.0651]
  FAS: Cycle 1 Day 1, Post-dose (n=52) | 0.02634 [0.0042 to 0.0846]
  FAS: Cycle 1 Day 15, 0 hours (n=48) | 0.03444 [0.0107 to 0.0735]
  FAS: Cycle 1 Day 15, Post-dose (n=46) | 0.03547 [0.0124 to 0.0882]
  FASLG: Cycle 1 Day 1, Baseline (n=55) | 0.00312 [0.0003 to 0.0281]
  FASLG: Cycle 1 Day 1, Post-dose (n=52) | 0.00343 [0.0004 to 0.0248]
  FASLG: Cycle 1 Day 15, 0 hours (n=48) | 0.00873 [0.0004 to 0.0338]
  FASLG: Cycle 1 Day 15, Post-dose (n=46) | 0.00820 [0.0005 to 0.0259]
  GAPDH: Cycle 1 Day 1, Baseline (n=55) | 0.77798 [0.3626 to 2.3473]
  GAPDH: Cycle 1 Day 1, Post-dose (n=52) | 0.74570 [0.3086 to 1.9921]
  GAPDH: Cycle 1 Day 15, 0 hours (n=48) | 0.46996 [0.3306 to 1.4609]
  GAPDH: Cycle 1 Day 15, Post-dose (n=46) | 0.43709 [0.2622 to 1.3683]
  GLI3: Cycle 1 Day 1, Baseline (n=35) | 0.00098 [0.0001 to 0.0101]
  GLI3: Cycle 1 Day 1, Post-dose (n=29) | 0.00107 [0.0001 to 0.0097]
  GLI3: Cycle 1 Day 15, 0 hours (n=10) | 0.00041 [0.0002 to 0.0051]
  GLI3: Cycle 1 Day 15, Post-dose (n=8) | 0.00054 [0.0004 to 0.0070]
  GSTA2: Cycle 1 Day 1, Baseline (n=22) | 0.00218 [0.0001 to 0.1397]
  GSTA2: Cycle 1 Day 1, Post-dose (n=6) | 0.00033 [0.0002 to 0.0086]
  GSTA2: Cycle 1 Day 15, Post-dose (n=2) | 0.00069 [0.0006 to 0.0008]
  GSTM1: Cycle 1 Day 1, Baseline (n=37) | 0.00958 [0.0007 to 0.0394]
  GSTM1: Cycle 1 Day 1, Post-dose (n=35) | 0.00885 [0.0009 to 0.0334]
  GSTM1: Cycle 1 Day 15, 0 hours (n=34) | 0.00706 [0.0004 to 0.0370]
  GSTM1: Cycle 1 Day 15, Post-dose (n=31) | 0.00642 [0.0004 to 0.0351]
  GSTM4: Cycle 1 Day 1, Baseline (n=54) | 0.00260 [0.0003 to 0.0132]
  GSTM4: Cycle 1 Day 1, Post-dose (n=50) | 0.00237 [0.0004 to 0.0134]
  GSTM4: Cycle 1 Day 15, 0 hours (n=47) | 0.00226 [0.0005 to 0.0091]
  GSTM4: Cycle 1 Day 15, Post-dose (n=44) | 0.00225 [0.0003 to 0.0098]
  GSTM5: Cycle 1 Day 1, Baseline (n=29) | 0.00045 [0.0000 to 0.0078]
  GSTM5: Cycle 1 Day 1, Post-dose (n=24) | 0.00050 [0.0000 to 0.0074]
  GSTM5: Cycle 1 Day 15, 0 hours (n=19) | 0.00065 [0.0001 to 0.0049]
  GSTM5: Cycle 1 Day 15, Post-dose (n=19) | 0.00094 [0.0002 to 0.0051]
  GSTP1: Cycle 1 Day 1, Baseline (n=55) | 0.28876 [0.0344 to 1.6475]
  GSTP1: Cycle 1 Day 1, Post-dose (n=52) | 0.28295 [0.0378 to 1.2982]
  GSTP1: Cycle 1 Day 15, 0 hours (n=48) | 0.19381 [0.0349 to 0.9610]
  GSTP1: Cycle 1 Day 15, Post-dose (n=46) | 0.19224 [0.0276 to 0.9227]
  GSTT1: Cycle 1 Day 1, Baseline (n=40) | 0.00061 [0.0000 to 0.0030]
  GSTT1: Cycle 1 Day 1, Post-dose (n=35) | 0.00065 [0.0001 to 0.0027]
  GSTT1: Cycle 1 Day 15, 0 hours (n=29) | 0.00064 [0.0002 to 0.0033]
  GSTT1: Cycle 1 Day 15, Post-dose (n=28) | 0.00066 [0.0002 to 0.0031]
  HRK: Cycle 1 Day 1, Baseline (n=48) | 0.00136 [0.0001 to 0.0635]
  HRK: Cycle 1 Day 1, Post-dose (n=41) | 0.00108 [0.0001 to 0.0526]
  HRK: Cycle 1 Day 15, 0 hours (n=11) | 0.00075 [0.0002 to 0.0041]
  HRK: Cycle 1 Day 15, Post-dose (n=13) | 0.00055 [0.0001 to 0.0060]
  IKZF1: Cycle 1 Day 1, Baseline (n=55) | 0.22553 [0.0053 to 0.6277]
  IKZF1: Cycle 1 Day 1, Post-dose (n=52) | 0.25975 [0.0204 to 0.5414]
  IKZF1: Cycle 1 Day 15, 0 hours (n=48) | 0.23670 [0.0072 to 0.5148]
  IKZF1: Cycle 1 Day 15, Post-dose (n=46) | 0.23925 [0.0072 to 0.5646]
  KMT2A: Cycle 1 Day 1, Baseline (n=55) | 0.03764 [0.0040 to 0.1704]
  KMT2A: Cycle 1 Day 1, Post-dose (n=52) | 0.03459 [0.0042 to 0.1663]
  KMT2A: Cycle 1 Day 15, 0 hours (n=48) | 0.02499 [0.0090 to 0.0708]
  KMT2A: Cycle 1 Day 15, Post-dose (n=46) | 0.02138 [0.0066 to 0.0844]
  KRT20: Cycle 1 Day 1, Baseline (n=2) | 0.00018 [0.0001 to 0.0002]
  LEF1: Cycle 1 Day 1, Baseline (n=55) | 0.18940 [0.0077 to 1.7280]
  LEF1: Cycle 1 Day 1, Post-dose (n=52) | 0.14479 [0.0089 to 1.6906]
  LEF1: Cycle 1 Day 15, 0 hours (n=48) | 0.07819 [0.0150 to 0.5602]
  LEF1: Cycle 1 Day 15, Post-dose (n=46) | 0.05586 [0.0121 to 0.8065]
  MCL1: Cycle 1 Day 1, Baseline (n=55) | 0.42021 [0.1390 to 1.0057]
  MCL1: Cycle 1 Day 1, Post-dose (n=52) | 0.44770 [0.1628 to 1.2938]
  MCL1: Cycle 1 Day 15, 0 hours (n=48) | 0.52160 [0.2694 to 1.4203]
  MCL1: Cycle 1 Day 15, Post-dose (n=46) | 0.61933 [0.2389 to 2.6947]
  MDC1: Cycle 1 Day 1, Baseline (n=55) | 0.01825 [0.0012 to 0.0535]
  MDC1: Cycle 1 Day 1, Post-dose (n=52) | 0.01825 [0.0012 to 0.0418]
  MDC1: Cycle 1 Day 15, 0 hours (n=48) | 0.01109 [0.0027 to 0.0346]
  MDC1: Cycle 1 Day 15, Post-dose (n=46) | 0.01034 [0.0022 to 0.0411]
  MRE11A: Cycle 1 Day 1, Baseline (n=55) | 0.00708 [0.0010 to 0.0210]
  MRE11A: Cycle 1 Day 1, Post-dose (n=52) | 0.00672 [0.0010 to 0.0277]
  MRE11A: Cycle 1 Day 15, 0 hours (n=48) | 0.00484 [0.0017 to 0.0109]
  MRE11A: Cycle 1 Day 15, Post-dose (n=46) | 0.00508 [0.0017 to 0.0147]
  MTOR: Cycle 1 Day 1, Baseline (n=55) | 0.01585 [0.0027 to 0.0498]
  MTOR: Cycle 1 Day 1, Post-dose (n=52) | 0.01636 [0.0029 to 0.0521]
  MTOR: Cycle 1 Day 15, 0 hours (n=48) | 0.01088 [0.0048 to 0.0288]
  MTOR: Cycle 1 Day 15, Post-dose (n=46) | 0.01122 [0.0041 to 0.0513]
  NHEJ1: Cycle 1 Day 1, Baseline (n=55) | 0.01162 [0.0026 to 0.0353]
  NHEJ1: Cycle 1 Day 1, Post-dose (n=52) | 0.01164 [0.0030 to 0.0352]
  NHEJ1: Cycle 1 Day 15, 0 hours (n=48) | 0.00974 [0.0040 to 0.0233]
  NHEJ1: Cycle 1 Day 15, Post-dose (n=46) | 0.01008 [0.0034 to 0.0271]
  NLRP2: Cycle 1 Day 1, Baseline (n=55) | 0.00237 [0.0002 to 0.0181]
  NLRP2: Cycle 1 Day 1, Post-dose (n=52) | 0.00226 [0.0004 to 0.0168]
  NLRP2: Cycle 1 Day 15, 0 hours (n=47) | 0.00301 [0.0002 to 0.0091]
  NLRP2: Cycle 1 Day 15, Post-dose (n=46) | 0.00283 [0.0002 to 0.0084]
  NOXA1: Cycle 1 Day 1, Baseline (n=52) | 0.00097 [0.0001 to 0.0079]
  NOXA1: Cycle 1 Day 1, Post-dose (n=48) | 0.00107 [0.0001 to 0.0069]
  NOXA1: Cycle 1 Day 15, 0 hours (n=43) | 0.00132 [0.0003 to 0.0032]
  NOXA1: Cycle 1 Day 15, Post-dose (n=42) | 0.00117 [0.0003 to 0.0032]
  PAX5: Cycle 1 Day 1, Baseline (n=55) | 0.05536 [0.0004 to 1.1631]
  PAX5: Cycle 1 Day 1, Post-dose (n=52) | 0.04433 [0.0007 to 0.8454]
  PAX5: Cycle 1 Day 15, 0 hours (n=30) | 0.00511 [0.0002 to 0.1024]
  PAX5: Cycle 1 Day 15, Post-dose (n=31) | 0.00369 [0.0001 to 0.2123]
  PDE4A: Cycle 1 Day 1, Baseline (n=55) | 0.00738 [0.0012 to 0.0578]
  PDE4A: Cycle 1 Day 1, Post-dose (n=52) | 0.00722 [0.0007 to 0.0566]
  PDE4A: Cycle 1 Day 15, 0 hours (n=48) | 0.00916 [0.0019 to 0.0202]
  PDE4A: Cycle 1 Day 15, Post-dose (n=46) | 0.00836 [0.0025 to 0.0235]
  PGK1: Cycle 1 Day 1, Baseline (n=55) | 0.19043 [0.1270 to 0.5490]
  PGK1: Cycle 1 Day 1, Post-dose (n=52) | 0.18772 [0.1103 to 0.5287]
  PGK1: Cycle 1 Day 15, 0 hours (n=48) | 0.14989 [0.0898 to 0.2804]
  PGK1: Cycle 1 Day 15, Post-dose (n=46) | 0.14783 [0.0649 to 0.2701]
  PIK3CA: Cycle 1 Day 1, Baseline (n=55) | 0.01664 [0.0057 to 0.0496]
  PIK3CA: Cycle 1 Day 1, Post-dose (n=52) | 0.01714 [0.0066 to 0.0535]
  PIK3CA: Cycle 1 Day 15, 0 hours (n=48) | 0.01154 [0.0068 to 0.0290]
  PIK3CA: Cycle 1 Day 15, Post-dose (n=46) | 0.01164 [0.0053 to 0.0273]
  PRKDC: Cycle 1 Day 1, Baseline (n=55) | 0.03206 [0.0023 to 0.1691]
  PRKDC: Cycle 1 Day 1, Post-dose (n=52) | 0.03543 [0.0023 to 0.1525]
  PRKDC: Cycle 1 Day 15, 0 hours (n=48) | 0.01964 [0.0049 to 0.0638]
  PRKDC: Cycle 1 Day 15, Post-dose (n=46) | 0.02159 [0.0051 to 0.0826]
  RAD50: Cycle 1 Day 1, Baseline (n=55) | 0.01482 [0.0017 to 0.0593]
  RAD50: Cycle 1 Day 1, Post-dose (n=52) | 0.01516 [0.0019 to 0.0525]
  RAD50: Cycle 1 Day 15, 0 hours (n=48) | 0.01129 [0.0041 to 0.0238]
  RAD50: Cycle 1 Day 15, Post-dose (n=46) | 0.01044 [0.0026 to 0.0244]
  RAD51: Cycle 1 Day 1, Baseline (n=54) | 0.00558 [0.0015 to 0.0484]
  RAD51: Cycle 1 Day 1, Post-dose (n=51) | 0.00573 [0.0010 to 0.0502]
  RAD51: Cycle 1 Day 15, 0 hours (n=47) | 0.00382 [0.0009 to 0.0222]
  RAD51: Cycle 1 Day 15, Post-dose (n=45) | 0.00356 [0.0004 to 0.0225]
  RAD52: Cycle 1 Day 1, Baseline (n=55) | 0.00384 [0.0007 to 0.0129]
  RAD52: Cycle 1 Day 1, Post-dose (n=52) | 0.00330 [0.0006 to 0.0115]
  RAD52: Cycle 1 Day 15, 0 hours (n=48) | 0.00221 [0.0008 to 0.0184]
  RAD52: Cycle 1 Day 15, Post-dose (n=46) | 0.00211 [0.0006 to 0.0085]
  RB1: Cycle 1 Day 1, Baseline (n=55) | 0.03434 [0.0050 to 0.1631]
  RB1: Cycle 1 Day 1, Post dose (n=52) | 0.03384 [0.0059 to 0.1365]
  RB1: Cycle 1 Day 15, 0 hours (n=48) | 0.01926 [0.0139 to 0.0579]
  RB1: Cycle 1 Day 15, Post-dose (n=46) | 0.01978 [0.0111 to 0.0887]
  RHEB: Cycle 1 Day 1, Baseline (n=55) | 0.02719 [0.0075 to 0.2452]
  RHEB: Cycle 1 Day 1, Post-dose (n=52) | 0.02287 [0.0078 to 0.1474]
  RHEB: Cycle 1 Day 15, 0 hours (n=48) | 0.01810 [0.0110 to 0.0377]
  RHEB: Cycle 1 Day 15, Post-dose (n=46) | 0.01835 [0.0107 to 0.0355]
  RPA1: Cycle 1 Day 1, Baseline (n=55) | 0.05178 [0.0097 to 0.1037]
  RPA1: Cycle 1 Day 1, Post-dose (n=52) | 0.05041 [0.0091 to 0.0897]
  RPA1: Cycle 1 Day 15, 0 hours (n=48) | 0.05348 [0.0262 to 0.1692]
  RPA1: Cycle 1 Day 15, Post-dose (n=46) | 0.05547 [0.0261 to 0.1925]
  SMAD1: Cycle 1 Day 1, Baseline (n=55) | 0.00858 [0.0001 to 0.1380]
  SMAD1: Cycle 1 Day 1, Post-dose (n=51) | 0.01116 [0.0003 to 0.1996]
  SMAD1: Cycle 1 Day 15, 0 hours (n=47) | 0.00167 [0.0004 to 0.0377]
  SMAD1: Cycle 1 Day 15, Post-dose (n=46) | 0.00197 [0.0004 to 0.0552]
  SYK: Cycle 1 Day 1, Baseline (n=55) | 0.06101 [0.0297 to 0.1445]
  SYK: Cycle 1 Day 1, Post-dose (n=52) | 0.05995 [0.0256 to 0.1346]
  SYK: Cycle 1 Day 15, 0 hours (n=48) | 0.04237 [0.0123 to 0.0918]
  SYK: Cycle 1 Day 15, Post-dose (n=46) | 0.04603 [0.0166 to 0.0979]
  TCF3: Cycle 1 Day 1, Baseline (n=55) | 0.09144 [0.0121 to 0.5337]
  TCF3: Cycle 1 Day 1, Post-dose (n=52) | 0.07770 [0.0138 to 0.4363]
  TCF3: Cycle 1 Day 15, 0 hours (n=48) | 0.04216 [0.0119 to 0.1552]
  TCF3: Cycle 1 Day 15, Post-dose (n=46) | 0.05154 [0.0126 to 0.2377]
  TNF: Cycle 1 Day 1, Baseline (n=55) | 0.00465 [0.0004 to 0.0335]
  TNF: Cycle 1 Day 1, Post-dose (n=52) | 0.00330 [0.0004 to 0.0262]
  TNF: Cycle 1 Day 15, 0 hours (n=48) | 0.00376 [0.0011 to 0.0230]
  TNF: Cycle 1 Day 15, Post-dose (n=46) | 0.00262 [0.0009 to 0.0170]
  TP53: Cycle 1 Day 1, Baseline (n=55) | 0.05412 [0.0013 to 0.3051]
  TP53: Cycle 1 Day 1, Post-dose (n=52) | 0.04778 [0.0020 to 0.2639]
  TP53: Cycle 1 Day 15, 0 hours (n=48) | 0.03196 [0.0085 to 0.0892]
  TP53: Cycle 1 Day 15, Post-dose (n=46) | 0.02741 [0.0052 to 0.0826]
  TP53BP1: Cycle 1 Day 1, Baseline (n=55) | 0.00386 [0.0005 to 0.0233]
  TP53BP1: Cycle 1 Day 1, Post-dose (n=52) | 0.00373 [0.0005 to 0.0214]
  TP53BP1: Cycle 1 Day 15, 0 hours (n=48) | 0.00205 [0.0009 to 0.0070]
  TP53BP1: Cycle 1 Day 15, Post-dose (n=46) | 0.00182 [0.0008 to 0.0098]
  VDAC3: Cycle 1 Day 1, Baseline (n=55) | 0.03899 [0.0095 to 0.1133]
  VDAC3: Cycle 1 Day 1, Post-dose (n=52) | 0.03701 [0.0114 to 0.1126]
  VDAC3: Cycle 1 Day 15, 0 hours (n=48) | 0.03748 [0.0192 to 0.0671]
  VDAC3: Cycle 1 Day 15, Post-dose (n=46) | 0.03621 [0.0189 to 0.0689]
  VPREB1: Cycle 1 Day 1, Baseline (n=52) | 0.08210 [0.0004 to 1.7113]
  VPREB1: Cycle 1 Day 1, Post-dose (n=47) | 0.08593 [0.0001 to 1.8106]
  VPREB1: Cycle 1 Day 15, 0 hours (n=25) | 0.00472 [0.0003 to 0.3317]
  VPREB1: Cycle 1 Day 15, Post-dose (n=28) | 0.00332 [0.0003 to 0.4981]
  XRCC2: Cycle 1 Day 1, Baseline (n=54) | 0.00260 [0.0002 to 0.0230]
  XRCC2: Cycle 1 Day 1, Post-dose (n=51) | 0.00297 [0.0003 to 0.0247]
  XRCC2: Cycle 1 Day 15, 0 hours (n=47) | 0.00125 [0.0003 to 0.0119]
  XRCC2: Cycle 1 Day 15, Post-dose (n=43) | 0.00124 [0.0003 to 0.0105]
  XRCC3: Cycle 1 Day 1, Baseline (n=55) | 0.00213 [0.0002 to 0.0143]
  XRCC3: Cycle 1 Day 1, Post-dose (n=50) | 0.00205 [0.0002 to 0.0127]
  XRCC3: Cycle 1 Day 15, 0 hours (n=46) | 0.00110 [0.0003 to 0.0048]
  XRCC3: Cycle 1 Day 15, Post-dose (n=43) | 0.00103 [0.0002 to 0.0065]
  XRCC4: Cycle 1 Day 1, Baseline (n=55) | 0.00175 [0.0004 to 0.0038]
  XRCC4: Cycle 1 Day 1, Post-dose (n=52) | 0.00183 [0.0004 to 0.0043]
  XRCC4: Cycle 1 Day 15, 0 hours (n=47) | 0.00172 [0.0004 to 0.0035]
  XRCC4: Cycle 1 Day 15, Post-dose (n=46) | 0.00179 [0.0006 to 0.0038]
  XRCC5: Cycle 1 Day 1, Baseline (n=55) | 0.22952 [0.0881 to 0.5646]
  XRCC5: Cycle 1 Day 15, 0 hours (n=48) | 0.18735 [0.1152 to 0.2920]
  XRCC5: Cycle 1 Day 15, Post-dose (n=46) | 0.17577 [0.1040 to 0.2685]
  XRCC6: Cycle 1 Day 1, Baseline (n=55) | 0.07688 [0.0117 to 0.2100]
  XRCC6: Cycle 1 Day 1, Post-dose (n=52) | 0.06620 [0.0109 to 0.1937]
  XRCC6: Cycle 1 Day 15, 0 hours (n=48) | 0.04898 [0.0163 to 0.1503]
  XRCC6: Cycle 1 Day 15, Post-dose (n=46) | 0.04495 [0.0126 to 0.1489]
  ZAP70: Cycle 1 Day 1, Baseline (n=55) | 0.11022 [0.0156 to 0.4971]
  ZAP70: Cycle 1 Day 1, Post-dose (n=52) | 0.10939 [0.0169 to 0.4442]
  ZAP70: Cycle 1 Day 15, 0 hours (n=48) | 0.18066 [0.0082 to 0.5237]
  ZAP70: Cycle 1 Day 15, Post-dose (n=46) | 0.15080 [0.0083 to 0.5991]
  XRCC5: Cycle 1 Day 1, Post-dose (n=52) | 0.22401 [0.0842 to 0.5260]

ADVERSE EVENTS:
Time Frame: AEs and SAEs were assessed from informed consent up to 28 calendar days after the last administration of investigational product, or up to the end of treatment visit (whichever is later) and to resolution/Grade 1 for treatment related AEs, up to 2 years.
Description: Events of veno-occlusive disease were reported up to 2 years after first dose of therapy. An event may appear as both an AE & SAE. However, what is presented are distinct events. An event may be categorized as serious in 1 participant & nonserious in another participant, or 1 participant may have experienced both a serious & nonserious event.
Arm/Group | Phase 1 - Dose-Finding: IV Inotuzumab Ozogamicin 1.2 mg/m^2 | Phase 1 - Dose-Finding: IV Inotuzumab Ozogamicin 1.6 mg/m^2 | Phase 1 - Dose-Finding: IV Inotuzumab Ozogamicin 1.8 mg/m^2 | Phase 1 - Expansion Phase: IV Inotuzumab Ozogamicin 1.8 mg/m^2 | Phase 2: IV Inotuzumab Ozogamicin 1.8mg/m^2
Serious Adverse Events (participants affected / at risk) | 3/3 | 4/12 | 8/9 | 10/13 | 26/35
Other Adverse Events (participants affected / at risk) | 3/3 | 12/12 | 9/9 | 10/13 | 34/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 - Dose-Finding: IV Inotuzumab Ozogamicin 1.2 mg/m^2 (N=3) | Phase 1 - Dose-Finding: IV Inotuzumab Ozogamicin 1.6 mg/m^2 (N=12) | Phase 1 - Dose-Finding: IV Inotuzumab Ozogamicin 1.8 mg/m^2 (N=9) | Phase 1 - Expansion Phase: IV Inotuzumab Ozogamicin 1.8 mg/m^2 (N=13) | Phase 2: IV Inotuzumab Ozogamicin 1.8mg/m^2 (N=35)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 1 | 5 | 8
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 2
Deafness (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Oral disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Disease progression (General disorders) | 0 | 1 | 0 | 1 | 3
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Venoocclusive liver disease (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 3
Abscess limb (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Enterococcal bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Necrotising fasciitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Periorbital cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 5
Pneumonia fungal (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pneumonia influenzal (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Septic shock (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Stenotrophomonas sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Central nervous system neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Neurological symptom (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 - Dose-Finding: IV Inotuzumab Ozogamicin 1.2 mg/m^2 (N=3) | Phase 1 - Dose-Finding: IV Inotuzumab Ozogamicin 1.6 mg/m^2 (N=12) | Phase 1 - Dose-Finding: IV Inotuzumab Ozogamicin 1.8 mg/m^2 (N=9) | Phase 1 - Expansion Phase: IV Inotuzumab Ozogamicin 1.8 mg/m^2 (N=13) | Phase 2: IV Inotuzumab Ozogamicin 1.8mg/m^2 (N=35)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 3 | 2 | 13
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 5
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0 | 8
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 2 | 6 | 3 | 7
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 4 | 5 | 2 | 19
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 3
External ear pain (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 1 | 0 | 0 | 2
Vision blurred (Eye disorders) | 0 | 0 | 1 | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 5 | 1 | 2 | 8
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 3 | 0 | 8
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 5 | 3 | 4 | 12
Oral disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 1
Retching (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 4 | 3 | 2 | 11
Asthenia (General disorders) | 1 | 1 | 0 | 0 | 2
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 1
Chills (General disorders) | 1 | 0 | 1 | 1 | 4
Facial pain (General disorders) | 0 | 0 | 1 | 0 | 1
Fatigue (General disorders) | 0 | 6 | 1 | 1 | 5
Generalised oedema (General disorders) | 0 | 0 | 1 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 2
Mucosal haemorrhage (General disorders) | 0 | 0 | 0 | 1 | 0
Oedema (General disorders) | 1 | 0 | 0 | 0 | 2
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0 | 3
Pain (General disorders) | 0 | 1 | 1 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 1 | 2 | 12
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1 | 1 | 9
Candida infection (Infections and infestations) | 0 | 0 | 1 | 0 | 3
Influenza (Infections and infestations) | 0 | 1 | 0 | 0 | 2
Otitis externa (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pseudomonal bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pulmonary mycosis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Septic shock (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Sinusitis fungal (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 4
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 2
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Activated partial thromboplastin time (Investigations) | 0 | 0 | 0 | 0 | 2
Alanine aminotransferase increased (Investigations) | 0 | 1 | 1 | 1 | 6
Aspartate aminotransferase increased (Investigations) | 0 | 3 | 5 | 3 | 8
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 4 | 1 | 7
Blood creatinine increased (Investigations) | 1 | 1 | 0 | 0 | 0
Blood test abnormal (Investigations) | 0 | 0 | 1 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 2 | 0 | 5 | 0 | 3
Lipase increased (Investigations) | 0 | 0 | 1 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 3
Weight increased (Investigations) | 0 | 0 | 2 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2 | 2 | 1 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 5
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 4
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 6
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 6
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 7
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 3
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 1 | 1 | 2
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 2 | 1 | 1 | 8
Nervous system disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 2
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 3
Paraesthesia (Nervous system disorders) | 0 | 0 | 2 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 2 | 0 | 4
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 2
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 2
Testicular pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1 | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 2
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1 | 3
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0 | 3
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1
Rash morbilliform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 1 | 2
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 5
Phlebitis (Vascular disorders) | 0 | 0 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 2
Lymph node pain (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Splenomegaly (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Catheter site erythema (General disorders) | 0 | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 1 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Transplant failure (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 60 days from the time submitted to the sponsor for review. The PI must remove any previously undisclosed Confidential Information (other than the Study results themselves) before public release.